CLINICAL TRIAL: NCT05267405
Title: Study on Disease Course and Quality of Life in Patients With Epilepsy (Mainz Epilepsy Registry)
Brief Title: Mainz Epilepsy Registry
Acronym: MAINZ-EPIREG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Dr. Yaroslav Winter, Head of Mainz Comprehensive Epilepsy and Sleep Medicine Center, Johannes Gutenberg University Mainz
Other Study IDs: MAINZ-EPIREG
Record Dates: First submitted 2022-02-11; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Epilepsy; Dissociative Seizures; Status Epilepticus
MeSH Terms: conditions — Epilepsy; Psychogenic Nonepileptic Seizures; Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no interventions, only observation — no interventions, only observation

SUMMARY:
Prospective longitudinal observational registry study of all patients with epilepsy treated in the Mainz Comprehensive Epilepsy and Sleep Medicine Center with the focus on the course of the disease and quality of life.

DETAILED DESCRIPTION:
Clinical parameters of patients, such as onset of the disease, prior medication, disease severity, which are important for the data analysis also collected retrospectively before the initiation of the registry. Data on the quality of life is collected only prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Epileptic or psychogenic seizures

Exclusion Criteria:

* age<18
* patients who cannot provide informed consent and don't have a legal guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated in Mainz Comprehensive Epilepsy and Sleep Medicine Center
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
monthly seizure frequency after 6 months | 6 months
  monthly seizure frequency at the follow-up after 6 months
European Quality of Life 5 dimensions Index (EQ 5D Index) | 6 months
  health-related quality of life measured by EQ5D-Index (European Quality of Life 5 dimensions), rating from 0 (worst possible state) to 1 (best possible state)
monthly seizure frequency after 12 months | 12 months
  monthly seizure frequency at the follow-up after 12 months
European Quality of Life 5 dimensions Index (EQ 5D Index) | 12 months
  health-related quality of life measured by EQ5D-Index (European Quality of Life 5 dimensions), rating from 0 (worst possible state) to 1 (best possible state)
Seizure freedom | 6 months
  percentage of patients without epileptic seizures
Seizure freedom | 12 months
  percentage of patients without epileptic seizures
interruption of status epilepticus | 48 hours
  percentage of patients with interrupted status epilepticus

SECONDARY OUTCOMES:
Resilience Scale 13 | 12 months
  Resilience Scale 13 (short version with 13 questions): 13-66 points correspond with low resilience, 67-72 with moderate and 73-91 with high resilience
Resilience Scale 13 | 24 months
  Resilience Scale 13 (short version with 13 questions): 13-66 points correspond with low resilience, 67-72 with moderate and 73-91 with high resilience
Multidimensional Fatigue Inventory | 12 months
  Multidimensional Fatigue Inventory: 20-item self-report instrument designed to measure fatigue. Measures range from 0-100, representing more severe fatigue at higher scores
Multidimensional Fatigue Inventory | 24 months
  Multidimensional Fatigue Inventory: 20-item self-report instrument designed to measure fatigue. Measures range from 0-100, representing more severe fatigue at higher scores
Beck Depression Inventory II | 12 months
  Beck Depression Inventory II: higher scores correspond to more severe depression (range 0-63)
Beck Depression Inventory II | 24 months
  Beck Depression Inventory II: higher scores correspond to more severe depression (range 0-63)
Berlin Social Support Scales (BSSS) | 12 months
  Berlin Social Support Scales (BSSS) is used to assess the amount of emotional, informational and instrumental support received by patients: Total scores ranged from 15 to 60, higher scores identify better support
Berlin Social Support Scales (BSSS) | 24 months
  Berlin Social Support Scales (BSSS) is used to assess the amount of emotional, informational and instrumental support received by patients: Total scores ranged from 15 to 60, higher scores identify better support
World Health Organization Quality of Life-BREF (WHOQOL-BREF) | 12 months
  World Health Organization Quality of Life-BREF (WHOQOL-BREF), a scale to assess overall quality of life with a range 0-100 (higher scores correspond better quality of life)
World Health Organization Quality of Life-BREF (WHOQOL-BREF) | 24 months
  World Health Organization Quality of Life-BREF (WHOQOL-BREF), a scale to assess overall quality of life with a range 0-100 (higher scores correspond better quality of life)
Pittsburgh Sleep Quality Index | 12 months
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances, scoring between 0 and 21 with higher scores corresponding to worse sleep quality
Pittsburgh Sleep Quality Index | 24 months
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances, scoring between 0 and 21 with higher scores corresponding to worse sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Yaroslav Winter, MD, MSc, Principal Investigator — Mainz Comprehensive Epilepsy and Sleep Medicine Center
Locations (1):
- Mainz Comprehensive Epilepsy and Sleep Medicine Center, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Winter Y, Abou Dargham R, Patino Tobon S, Groppa S, Fuest S. Cenobamate as an Early Adjunctive Treatment in Drug-Resistant Focal-Onset Seizures: An Observational Cohort Study. CNS Drugs. 2024 Sep;38(9):733-742. doi: 10.1007/s40263-024-01109-9. Epub 2024 Aug 3. PMID 39096467
- [Derived] Winter Y, Sandner K, Vieth T, Gonzalez-Escamilla G, Stuckrad-Barre SV, Groppa S. Third-Generation Antiseizure Medication in the Treatment of Benzodiazepine-Refractory Status Epilepticus in Poststroke Epilepsy: A Retrospective Observational Register-Based Study. CNS Drugs. 2023 Oct;37(10):929-936. doi: 10.1007/s40263-023-01039-y. Epub 2023 Oct 2. PMID 37784006